CLINICAL TRIAL: NCT03652597
Title: Neuro-Cardiac-Guided Transcranial Magnetic Stimulation: a Method to Probe the Depression Network. Replication and Dose-response
Brief Title: Neuro-Cardiac-Guided Transcranial Magnetic Stimulation: Replication and Dose-response.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utrecht University (Other)
Collaborators: Research institute Brainclinics (Unknown)
Responsible Party: Principal Investigator, Tabitha Iseger, Principal investigator, Utrecht University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NL63092.041.17
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
Keywords: Target engagement; TMS; Heart-brain pathway; Depression; Neuromodulation; DLPFC; Heart rate
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left (Active Comparator): Subjects are ascribed to left hemispheric stimulation
  Interventions: Device: Transcranial magnetic stimulation (TMS)
- Right (Active Comparator): Subjects are ascribed to right hemispheric stimulation
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — Subjects receive TMS on several cortical brain locations, while recording the heart rate.

SUMMARY:
Autonomic regulation is disturbed in patients with major depressive disorder (MDD), indicated by a higher heart rate (HR) and lower heart rate variability (HRV). Moreover, the heart seems to be functionally connected via the vagus nerve (VN) to other brain structures that are dysregulated in depression, such as the subgenual anterior cingulate cortex (sgACC), and the dorsolateral prefrontal cortex (DLPFC), suggesting dysregulated network function in MDD. In line with this network dysregulation hypothesis of MDD, optimal transcranial magnetic stimulation (TMS) sites are currently thought to be those that show functional connectivity to the sgACC such as the DLPFC and multiple studies have shown that stimulation of the DLPFC, sgACC and nervus vagus decreased heart rate, suggestive of parasymphatetic action. It is hypothesized that this influence on parasympathetic activity can be used as a functional outcome measure reflecting adequate targeting of the DLPFC-sgACC network, similar to the motor evoked potential (MEP) as functional key measure for primary motor cortex stimulation. Recently, a pilot study was conducted, proposing a new functional neuronavigation method for localizing the frontal area representation of DLPFC-sgACC connectivity using HR, called: Neuro-Cardiac-Guided TMS (NCG-TMS), which is being replicated in the current study. .

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Between ages 18-60

Exclusion Criteria:

* No prior experience with epilepsy
* No pregnancy
* No metal in the head
* No cochlear implants

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
Heart rate during stimulation, converted to RR intervals | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Arns, Phd., Study Director — Research institute Brainclinics
Locations (1):
- Research institute Brainclinics, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No